CLINICAL TRIAL: NCT01040793
Title: Randomised, Double-blind, Placebo-controlled, 3-way Cross-over Study to Determine the Effect of Treatment of Orally Inhaled BI 1744 CL (5 µg [2 Actuations of 2.5 µg] and 10 µg [2 Actuations of 5 µg]) Delivered by the Respimat® Inhaler on Exercise Endurance Time During Constant Work Rate Cycle Ergometry in Patients With Chronic Obstructive Pulmonary Disease.
Brief Title: Effect of Treatment BI 1744 CL (5 and 10 mcg) Versus Placebo on Exercise Endurance Time During Constant Work Rate Cycle Ergometry II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1222.38; 2009-014416-35 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-12-29; First posted 2009-12-30 (Estimated); Results first posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — olodaterol

ARMS (3):
- Olodaterol (BI 1744) Low (Experimental): Low dose inhaled orally once daily from the Respimat inhaler
  Interventions: Drug: Olodaterol (BI 1744); Drug: Olodaterol (BI1744); Drug: Olodaterol (BI 1744) placebo
- Olodaterol (BI 1744) High (Experimental): High dose inhaled orally once daily from the Respimat inhaler
  Interventions: Drug: Olodaterol (BI 1744)
- Placebo (Placebo Comparator): Olodaterol (BI 1744) placebo inhaled orally from the Respimat inhaler
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olodaterol (BI 1744) — Comparison of low and high dose on exercise endurance time in COPD patients
  Arms: Olodaterol (BI 1744) Low
Drug: Olodaterol (BI 1744) — Comparison of low and high dose on exercise endurance time in COPD patients
  Arms: Olodaterol (BI 1744) High
Drug: Placebo — Comparison of low and high dose and placebo on exercise endurance time in COPD patients
  Arms: Placebo
Drug: Olodaterol (BI1744) — Comparison of low and high dose on exercise endurance time in COPD patients
  Arms: Olodaterol (BI 1744) Low
Drug: Olodaterol (BI 1744) placebo — Placebo that represents olodaterol
  Arms: Olodaterol (BI 1744) Low

SUMMARY:
To compare the effects of BI 1744 CL versus placebo on exercise tolerance after 6 weeks of treatment in patients with Chronic Obstructive Pulmonary Disease.

ELIGIBILITY:
Inclusion criteria:

1. Signed informed consent prior to participation.
2. Diagnosis of chronic obstructive pulmonary disease and post-bronchodilator FEV1(Forced Expiratory Volume in 1 sec) <80% of predicted normal and post-bronchodilator FEV1(Forced Expiratory Volume in 1 sec)/FVC of < 70% at Visit 1.
3. Male or female between 40 and 75 years of age.
4. Current or ex-smokers with smoking history of more than 10-pack years.
5. Able to perform technically acceptable pulmonary function tests, multiple exercise tests and able to maintain records.
6. Able to inhale medication in a competent manner from a metered-dose inhaler and Respimat inhaler.

Exclusion criteria:

1. Patients with clinically relevant abnormal baseline haematology, blood chemistry, or urinalysis; all patients with an SGOT >x2 ULN, SGPT >x2 ULN, bilirubin >x2 ULN or creatinine >x2 ULN.
2. Patients with a history of asthma and/or total blood eosinophil count of 600 cells/mm3.
3. Patients with thyrotoxicosis, paroxysmal tachycardia (>100 beats per minute).
4. Patients with a history of myocardial infarction within 1 year of screening visit, unstable or life-threatening cardiac arrhythmia, hospitalization for heart failure within the past year, known active tuberculosis, a malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years, life-threatening pulmonary obstruction, cystic fibrosis, clinically evident bronchiectasis, significant alcohol or drug abuse or contraindications to exercise.
5. Patients who have undergone thoracotomy with pulmonary resection.
6. Patients being treated with oral beta-adrenergics or oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day.
7. Patients who regularly use daytime oxygen for more than one hour per day.
8. Patients who have completed a pulmonary rehabilitation program in the six weeks prior to the screening visit or patients who are currently in a pulmonary rehabilitation program.
9. Patients who have a limitation of exercise performance as a result of factors other than fatigue or exertional dyspnea.
10. Pregnant or nursing women.
11. Women of childbearing potential not using two effective methods of birth control (one barrier and one non-barrier).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2010-01; Primary Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (19):
- Austria (2):
  - 1222.38.4380 Boehringer Ingelheim Investigational Site, Hallein
  - 1222.38.4381 Boehringer Ingelheim Investigational Site, Leoben
- Belgium (4):
  - 1222.38.32004 Boehringer Ingelheim Investigational Site, Brussels
  - 1222.38.32002 Boehringer Ingelheim Investigational Site, Edegem
  - 1222.38.32001 Boehringer Ingelheim Investigational Site, Leuven
  - 1222.38.32003 Boehringer Ingelheim Investigational Site, Liège
- Canada (4):
  - 1222.38.1082 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1222.38.1081 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1222.38.1083 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1222.38.1080 Boehringer Ingelheim Investigational Site, Montreal, Quebec
- Germany (6):
  - 1222.38.4980 Boehringer Ingelheim Investigational Site, Berlin
  - 1222.38.4985 Boehringer Ingelheim Investigational Site, Cologne
  - 1222.38.4983 Boehringer Ingelheim Investigational Site, Dortmund
  - 1222.38.4984 Boehringer Ingelheim Investigational Site, Großhansdorf
  - 1222.38.4981 Boehringer Ingelheim Investigational Site, Kiel
  - 1222.38.4986 Boehringer Ingelheim Investigational Site, Koblenz
- Russia (3):
  - 1222.38.7080 Boehringer Ingelheim Investigational Site, Moscow
  - 1222.38.7081 Boehringer Ingelheim Investigational Site, Moscow
  - 1222.38.7082 Boehringer Ingelheim Investigational Site, Saint Petersburg

REFERENCES:
- [Derived] Maltais F, Kirsten AM, Hamilton A, De Sousa D, Voss F, Decramer M. Evaluation of the effects of olodaterol on exercise endurance in patients with chronic obstructive pulmonary disease: results from two 6-week crossover studies. Respir Res. 2016 Jul 6;17(1):77. doi: 10.1186/s12931-016-0389-5. PMID 27383762

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomised, double-blind, placebo-controlled, 3-way crossover trial. The duration of each treatment period was 6 weeks with a 14 day washout period between treatments.
Groups:
- Placebo / Olo 5mcg / Olo 10mcg: Patients were administered placebo in the first period, Olodaterol 5 mcg qd in the second period and Olodaterol 10 mcg qd in the third period. Olodaterol was administered via the Respimat inhaler.
- Placebo / Olo 10mcg / Olo 5mcg: Patients were administered placebo in the first period, Olodaterol 10 mcg qd in the second period and Olodaterol 5 mcg qd in the third period. Olodaterol was administered via the Respimat inhaler.
- Olo 5mcg/ Placebo / Olo 10mcg: Patients were administered Olodaterol 5 mcg qd in the first period, placebo in the second period and Olodaterol 10 mcg qd in the third period. Olodaterol was administered via the Respimat inhaler.
- Olo 5mcg / Olo 10mcg / Placebo: Patients were administered Olodaterol 5 mcg qd in the first period, Olodaterol 10 mcg qd in the second period and placebo in the third period. Olodaterol was administered via the Respimat inhaler.
- Olo 10mcg / Placebo / Olo 5mcg: Patients were administered Olodaterol 10 mcg qd in the first period, placebo in the second period and Olodaterol 5 mcg qd in the third period. Olodaterol was administered via the Respimat inhaler.
- Olo 10mcg / Olo 5mcg / Placebo: Patients were administered Olodaterol 10 mcg qd in the first period, Olodaterol 5 mcg qd in the second period and placebo in the third period. Olodaterol was administered via the Respimat inhaler.
Period: Overall Study
Arm/Group | Placebo / Olo 5mcg / Olo 10mcg | Placebo / Olo 10mcg / Olo 5mcg | Olo 5mcg/ Placebo / Olo 10mcg | Olo 5mcg / Olo 10mcg / Placebo | Olo 10mcg / Placebo / Olo 5mcg | Olo 10mcg / Olo 5mcg / Placebo
Started | 26 (Entered and treated) | 26 | 26 | 26 | 26 | 27
Completed | 20 | 21 | 23 | 22 | 22 | 26
Not Completed | 6 | 5 | 3 | 4 | 4 | 1
Not completed — Adverse Event | 5 | 3 | 0 | 2 | 2 | 1
Not completed — Protocol Violation | 1 | 1 | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Other reasons not listed above | 0 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Total number of patients treated in the study. This was a randomised, double-blind, placebo-controlled, 3-way crossover trial. 151 patients were assigned randomly to one of 3 treatment sequences in which they received each of 3 treatments. The duration of each treatment period was 6 weeks with a 14 day washout period between treatments.
Arm/Group | Overall Study
Number analyzed (Participants) | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 116

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Endurance Time After 6 Weeks
Description: Primary endpoint was endurance time during constant work rate ergometry to symptom limitation at 75% of maximal work capacity after 6 weeks of treatment. Mixed effects model on log10 transformation data. Adjusted means are back transformed to report as geometric means. Standard errors (SEs) are calculated using the delta method.
Time Frame: 6 weeks
Population: Full analysis set (FAS). FAS is defined as all patients that were randomised, received treatment and had baseline data and any evaluable post-dose data for the primary endpoint.
Measure: Geometric Mean (Standard Error); unit: seconds
Groups:
- Placebo: Matching Placebo delivered by the Respimat Inhaler.
- Olo 5 mcg qd: Olodaterol 5 mcg qd delivered by the Respimat Inhaler.
- Olo 10 mcg qd: Olodaterol 10 mcg qd delivered by the Respimat Inhaler.
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 146 | 141 | 140
seconds | 354.33 (12.069) | 396.31 (13.680) | 391.45 (13.566)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0018, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline endurance time and period as fixed and patient as random effect. Means, CI back-transformed; Ratio to placebo = 1.118, 95% CI [1.043 to 1.199], Standard Error of Mean 0.040 — Olo 5 mcg divided by Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0052, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Ratio to placebo = 1.105, 95% CI [1.030 to 1.184], Standard Error of Mean 0.039 — Olo 10 mcg divided by Placebo

2. Secondary Outcome: Adjusted Mean Inspiratory Capacity at Isotime After 6 Weeks
Description: Isotime is defined as the endurance time of the constant work rate exercise test of shortest duration from Baseline visit, and Week 6 of each of the three treatment periods.
Time Frame: 6 weeks
Population: Full analysis set (FAS). FAS is defined as all patients that were randomised, received treatment and had baseline data and any evaluable post-dose data for the primary endpoint. Only patients who have baseline and at least one post-baseline measurement available were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 146 | 141 | 139
liters | 2.162 (0.039) | 2.246 (0.039) | 2.328 (0.039)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0155, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.084, 95% CI [0.016 to 0.152], Standard Error of Mean 0.035 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.166, 95% CI [0.098 to 0.234], Standard Error of Mean 0.034 — Olo 10 mcg minus Placebo

3. Secondary Outcome: Adjusted Mean Borg Scale of Breathing Discomfort at Isotime After 6 Weeks
Description: Isotime is defined as the endurance time of the constant work rate exercise test of shortest duration from Baseline visit, and Week 6 of each of the three treatment periods.
  Borg scale rates discomfort with breathing at rest, during exercise and at end-exercise on a scale from 0=Nothing at all to 10=Maximal discomfort.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 146 | 141 | 140
Scores on a scale | 5.585 (0.177) | 5.250 (0.180) | 5.520 (0.181)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.1176, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = -0.366, 95% CI [-0.757 to 0.085], Standard Error of Mean 0.214 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.7591, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = -0.066, 95% CI [-0.486 to 0.355], Standard Error of Mean 0.214 — Olo 10 mcg minus Placebo

4. Secondary Outcome: Adjusted Mean Inspiratory Capacity at Pre-exercise After 6 Weeks
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 146 | 141 | 138
liters | 2.273 (0.036) | 2.437 (0.036) | 2.468 (0.037)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.164, 95% CI [0.094 to 0.234], Standard Error of Mean 0.036 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.195, 95% CI [0.125 to 0.265], Standard Error of Mean 0.036 — Olo 10 mcg minus Placebo

5. Secondary Outcome: Adjusted Mean Inspiratory Capacity at End of Exercise After 6 Weeks
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 146 | 141 | 139
liters | 2.158 (0.039) | 2.236 (0.040) | 2.330 (0.040)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0245, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.078, 95% CI [0.010 to 0.146], Standard Error of Mean 0.034 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.172, 95% CI [0.105 to 0.240], Standard Error of Mean 0.034 — Olo 10 mcg minus Placebo

6. Secondary Outcome: Adjusted Mean Borg Scale of Breathing Discomfort at Pre-exercise After 6 Weeks
Description: Borg scale rates discomfort with breathing at rest, during exercise and at end-exercise on a scale from 0=Nothing at all to 10=Maximal discomfort.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 146 | 141 | 140
Scores on a scale | 0.389 (0.062) | 0.315 (0.063) | 0.364 (0.064)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.2897, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = -0.074, 95% CI [-0.211 to 0.063], Standard Error of Mean 0.070 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.7199, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = -0.025, 95% CI [-0.162 to 0.112], Standard Error of Mean 0.069 — Olo 10 mcg minus Placebo

7. Secondary Outcome: Adjusted Mean Borg Scale of Breathing Discomfort at End of Exercise After 6 Weeks
Description: as for outcome 6
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 146 | 141 | 140
Scores on a scale | 7.010 (0.129) | 7.101 (0.131) | 7.351 (0.132)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.5313, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.091, 95% CI [-0.196 to 0.379], Standard Error of Mean 0.146 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0198, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.341, 95% CI [0.055 to 0.628], Standard Error of Mean 0.146 — Olo 10 mcg minus Placebo

8. Secondary Outcome: Adjusted Mean Functional Residual Capacity 30 Minutes Pre-dose After 6 Weeks
Description: Measured using body plethysmography
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 147 | 145 | 141
liters | 4.842 (0.062) | 4.757 (0.063) | 4.723 (0.063)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.1048, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = -0.086, 95% CI [-0.190 to 0.018], Standard Error of Mean 0.053 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0246, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = -0.120, 95% CI [-0.224 to -0.015], Standard Error of Mean 0.053 — Olo 10 mcg minus Placebo

9. Secondary Outcome: Adjusted Mean Functional Residual Capacity 1 Hour Post-dose After 6 Weeks
Description: Measured using body plethysmography
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 147 | 145 | 141
liters | 4.770 (0.065) | 4.557 (0.065) | 4.583 (0.065)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = -0.213, 95% CI [-0.318 to -0.108], Standard Error of Mean 0.053 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = -0.187, 95% CI [-0.293 to -0.082], Standard Error of Mean 0.054 — Olo 10 mcg minus Placebo

10. Secondary Outcome: Adjusted Mean Inspiratory Capacity 30 Minutes Pre-dose After 6 Weeks
Description: Measured using body plethysmography
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 147 | 146 | 142
liters | 2.463 (0.041) | 2.613 (0.041) | 2.618 (0.042)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.150, 95% CI [0.071 to 0.228], Standard Error of Mean 0.040 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.154, 95% CI [0.076 to 0.233], Standard Error of Mean 0.040 — Olo 10 mcg minus Placebo

11. Secondary Outcome: Adjusted Mean Inspiratory Capacity 1 Hour Post-dose After 6 Weeks
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 147 | 146 | 142
liters | 2.493 (0.040) | 2.725 (0.040) | 2.696 (0.040)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.232, 95% CI [0.162 to 0.303], Standard Error of Mean 0.036 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.203, 95% CI [0.133 to 0.273], Standard Error of Mean 0.036 — Olo 10 mcg minus Placebo

12. Secondary Outcome: Adjusted Mean Total Lung Capacity 30 Minutes Pre-dose After 6 Weeks
Description: Measured using body plethysmography
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 147 | 146 | 142
liters | 7.311 (0.067) | 7.368 (0.067) | 7.340 (0.068)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.3109, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.057, 95% CI [-0.053 to 0.166], Standard Error of Mean 0.056 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.6080, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.029, 95% CI [-0.081 to 0.138], Standard Error of Mean 0.056 — Olo 10 mcg minus Placebo

13. Secondary Outcome: Adjusted Mean Total Lung Capacity 1 Hour Post-dose After 6 Weeks
Description: Measured using body plethysmography
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 147 | 146 | 142
liters | 7.262 (0.069) | 7.285 (0.069) | 7.272 (0.069)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.6809, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.023, 95% CI [-0.087 to 0.133], Standard Error of Mean 0.056 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.8580, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.010, 95% CI [-0.100 to 0.120], Standard Error of Mean 0.056 — Olo 10 mcg minus Placebo

14. Secondary Outcome: Adjusted Mean Forced Expiratory Volume in 1 Second, 30 Minutes Pre-dose After 6 Weeks
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 146 | 143 | 139
liters | 1.520 (0.024) | 1.630 (0.025) | 1.630 (0.025)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.110, 95% CI [0.073 to 0.148], Standard Error of Mean 0.019 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.110, 95% CI [0.073 to 0.148], Standard Error of Mean 0.019 — Olo 10 mcg minus Placebo

15. Secondary Outcome: Adjusted Mean Forced Expiratory Volume in 1 Second, 1 Hour Post-dose After 6 Weeks
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 146 | 143 | 139
liters | 1.577 (0.026) | 1.768 (0.026) | 1.771 (0.026)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.192, 95% CI [0.151 to 0.233], Standard Error of Mean 0.021 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.195, 95% CI [0.153 to 0.236], Standard Error of Mean 0.021 — Olo 10 mcg minus Placebo

16. Secondary Outcome: Adjusted Mean Forced Vital Capacity, 30 Minutes Pre-dose After 6 Weeks
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 146 | 143 | 139
liters | 3.103 (0.039) | 3.222 (0.040) | 3.222 (0.040)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p = 0.0013, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.119, 95% CI [0.047 to 0.191], Standard Error of Mean 0.036 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p = 0.0013, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.119, 95% CI [0.047 to 0.191], Standard Error of Mean 0.037 — Olo 10 mcg minus Placebo

17. Secondary Outcome: Adjusted Mean Forced Vital Capacity, 1 Hour Post-dose After 6 Weeks
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 146 | 143 | 139
liters | 3.144 (0.039) | 3.409 (0.040) | 3.425 (0.040)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.265, 95% CI [0.196 to 0.333], Standard Error of Mean 0.035 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.281, 95% CI [0.212 to 0.350], Standard Error of Mean 0.035 — Olo 10 mcg minus Placebo

18. Secondary Outcome: Adjusted Mean Peak Expiratory Flow Rate, 30 Minutes Pre-dose After 6 Weeks
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters/second
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 146 | 143 | 139
liters/second | 4.258 (0.081) | 4.539 (0.081) | 4.549 (0.082)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.281, 95% CI [0.156 to 0.405], Standard Error of Mean 0.063 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.291, 95% CI [0.166 to 0.416], Standard Error of Mean 0.063 — Olo 10 mcg minus Placebo

19. Secondary Outcome: Adjusted Mean Peak Expiratory Flow Rate, 1 Hour Post-dose After 6 Weeks
Time Frame: 6 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters/second
Arm/Group | Placebo | Olo 5 mcg qd | Olo 10 mcg qd
Number analyzed (Participants) | 146 | 143 | 139
liters/second | 4.324 (0.085) | 4.904 (0.085) | 4.876 (0.086)
Statistical Analysis 1: Comparison: Placebo vs Olo 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.580, 95% CI [0.441 to 0.719], Standard Error of Mean 0.070 — Olo 5 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olo 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed effects repeated measures with treatment, baseline and period as fixed and patient as random effect; Mean Difference (Final Values) = 0.552, 95% CI [0.412 to 0.691], Standard Error of Mean 0.071 — Olo 10 mcg minus Placebo

20. Secondary Outcome: Change From Baseline to Day 43 in Blood Pressure
Description: Change from Baseline to Day 43 in Blood Pressure with spirometry. Baseline is defined as mean of pre-treatment values at a given time point.
Time Frame: Baseline and Week 6
Population: Treated set. Statistics only include patients with both a baseline and a post dose value.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Olo 5 mcg: Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 10 mcg: Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler.
Arm/Group | Placebo | Olo 5 mcg | Olo 10 mcg
Number analyzed (Participants) | 147 | 144 | 139
mmHg
  Systolic blood pressure | -0.5 (15.87) | -1.5 (15.47) | -1.4 (15.31)
  Diastolic blood pressure | -0.8 (8.95) | -1.8 (8.35) | -2.2 (9.5)

21. Secondary Outcome: Change From Baseline to Day 43 in Pulse Rate
Description: Change from Baseline to Day 43 in Pulse rate with spirometry. Baseline is defined as mean of pre-treatment values at a given time point.
Time Frame: Baseline and Week 6
Population: Treated set. Statistics only include patients with both a baseline and a post dose value.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | Olo 5 mcg | Olo 10 mcg
Number analyzed (Participants) | 147 | 144 | 139
beats/min | -2.3 (12.33) | -1.8 (11.69) | -1.6 (10.36)

22. Secondary Outcome: Number of Patients With Notable Changes in Heart Rate
Description: Number of Patients with notable changes in heart rate (HR). Notable HR increase defined as >=25% increase and on-treatment HR > 100 bpm; Notable HR decrease defined as >=25% decrease and on-treatment HR < 50 bpm.
Time Frame: Baseline and Week 6
Population: Treated set.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Olo 5 mcg | Olo 10 mcg
Number analyzed (Participants) | 147 | 143 | 140
percentage of participants
  30 min pre-dose: increase | 0.7 | 0.7 | 0.0
  30 min pre-dose: decrease | 0.7 | 1.4 | 2.9
  30 min pre-dose: no notable change | 98.6 | 97.9 | 97.1
  40 min post-dose: increase (N=147,142,140) | 0.0 | 0.0 | 0.0
  40 min post-dose: decrease (N=147,142,140) | 0.7 | 4.2 | 3.6
  40 min post-dose: no notable change(N=147,142,140) | 99.3 | 95.8 | 96.4

23. Secondary Outcome: Number of Patients With Notable Increase in PR Intervals
Description: Number of Patients with notable increase in PR intervals. Notable PR interval increase defined as >=25% increase and on-treatment PR interval > 200 ms.
Time Frame: Baseline and Week 6
Population: Treated set.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Olo 5 mcg | Olo 10 mcg
Number analyzed (Participants) | 147 | 143 | 140
percentage of participants
  30 min pre-dose: increase | 0.0 | 0.0 | 0.0
  30 min pre-dose: no increase | 100.0 | 100.0 | 100.0
  40 min post-dose: increase (N=147, 142, 140) | 0.7 | 0.0 | 0.0
  40 min post-dose: no increase (N=147, 142, 140) | 99.3 | 100.0 | 100.0

24. Secondary Outcome: Number of Patients With Notable Increase in QRS Intervals
Description: Number of Patients with notable increase in QRS intervals. Notable QRS interval increase defined as >=10% increase and on-treatment QRS interval > 110 ms.
Time Frame: Baseline and Week 6
Population: Treated set.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Olo 5 mcg | Olo 10 mcg
Number analyzed (Participants) | 147 | 143 | 140
percentage of participants
  30 min pre-dose: increase | 0.7 | 0.7 | 0.7
  30 min pre-dose: no increase | 99.3 | 99.3 | 99.3
  40 min post-dose: increase (N=147, 142, 140) | 1.4 | 0.7 | 0.7
  40 min post-dose: no increase (N=147, 142, 140) | 98.6 | 99.3 | 99.3

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- Placebo: Matching Placebo delivered by the Respimat resp. Aerolizer Inhaler.
Arm/Group | Placebo | Olo 5 mcg | Olo 10 mcg
Serious Adverse Events (participants affected / at risk) | 3/149 | 8/150 | 3/147
Other Adverse Events (participants affected / at risk) | 9/149 | 8/150 | 4/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=149) | Olo 5 mcg (N=150) | Olo 10 mcg (N=147)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Foreign body aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=149) | Olo 5 mcg (N=150) | Olo 10 mcg (N=147)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 | 8 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication